CLINICAL TRIAL: NCT00109005
Title: A Randomized Phase II Study of Oral Lenalidomide (Revlimid [TM]), an Antiangiogenic and Immunomodulatory Agent, in Subjects With Stage IV Ocular Melanoma
Brief Title: Lenalidomide (Revlimid) to Treat Advanced Ocular Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Caryn Steakley, R.N., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 050095; 05-C-0095; NCT00112606 (obsolete NCT alias)
Record Dates: First submitted 2005-04-21; First posted 2005-04-22 (Estimated); Results first posted 2012-10-30 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-11

CONDITIONS: Melanoma
Keywords: Response Rate; Toxicity; Progression-Free Survival; Overall Survival; Pharmacokinetic; Ocular Melanoma
MeSH Terms: conditions — Melanoma; Uveal Melanoma | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 - 25 mg lenalidomide (Revlimid) (Experimental): oral dose (1 capsule) lenalidomide 25 mg per day 7 days a week for 3 weeks
  Interventions: Drug: Revlimid
- Cohort 2 - 5 mg lenalidomide (Revlimid) (Experimental): oral dose (1 capsule) lenalidomide 5 mg per day 7 days a week for 3 weeks
  Interventions: Drug: Revlimid

INTERVENTIONS:
Drug: Revlimid — oral dose (1 capsule) 25 mg per day 7 days a week for cohort 1 oral dose (1 capsule) 5 mg per day 7 days a week for cohort 2
  Other Names: Lenalidomide

SUMMARY:
This study will test whether an experimental drug called Revlimid (lenalidomide) can reduce tumor size and prolong survival in patients with metastatic melanoma (melanoma that has spread beyond the original tumor site). It will also examine the toxicity and blood effects of Revlimid.

Patients 18 years of age and older with stage IV ocular melanoma may be eligible for this study. Candidates are screened with a medical history and physical and examination, blood and urine tests, electrocardiogram, chest x-ray, computed tomography (CT) scan and other imaging scans if needed, such as a bone scan, magnetic resonance imaging (MRI), ultrasound, or positron emission tomography (PET).

Participants are admitted to the National Institutes of Health (NIH) Clinical Center for 24 hours for their first oral dose of Revlimid. During the hospital stay, blood is drawn before the dose is given and again at 0.25, 0.5, 1, 2, 4, 6, 9, 12 and 24 hours after dosing to see how the body handles the drug. If the drug is well tolerated, patients are sent home with a 21-day supply of drug to take once a day for 21 days, then go off drug 7 days. This regimen constitutes one 28-day treatment cycle. Treatment cycles may continue for up to 2 years.

Patients keep a daily diary of side effects and have blood drawn once a week. The drug dose may be adjusted according to the laboratory test results. If unacceptable toxicity occurs, treatment may be stopped.

Patients who agree to be biopsied undergo this procedure before treatment begins and at the end of treatment cycles 3 and 6. A small area of skin is numbed with medicine and a small piece of tumor is removed with a needle or by a small cut in the tumor. The tissue is examined under a microscope.

Patients return to NIH after the first month of treatment and then every 3 months to evaluate their tumors and treatment of side effects. The visits include a physical examination, x-rays and scans to evaluate tumors. Visits are scheduled every 3 months while on treatment; then every 3 months for 2 years afterwards; then every 4 months for 1 year; and as needed after that. Patients will have a brain magnetic resonance imaging scan once a year to watch for new tumor areas.

DETAILED DESCRIPTION:
Background:

* Patients with stage IV ocular melanoma have very few available treatment options and an overall poor prognosis.
* Pre-clinical and early clinical evidence suggest that lenalidomide has activity against solid tumors.
* This trial is designed to evaluate the safety and efficacy of two different doses of a novel antiangiogenic and immunomodulatory agent, lenalidomide (Revlimid ).

Objectives:

Primary Objectives:

* Determine the response rate to lenalidomide at two dose levels for patients with Stage IV ocular melanoma.
* To determine the toxicity of lenalidomide at two dose levels in this setting.

Secondary Objectives:

* To determine the progression free and overall survival of patients with Stage IV ocular melanoma treated with lenalidomide.
* When easily accessible, obtain tissue at baseline and during therapy to evaluate the effects of these agents on pathways, thought to be modulated by lenalidomide in pre-clinical studies.
* To determine the pharmacokinetics of lenalidomide at these two doses in patients with Stage IV ocular melanoma.
* To determine if there is a dose level with potentially superior efficacy and acceptable toxicity.

Eligibility:

* Patients > 18 years of age with stage IV ocular melanoma, who have measurable disease.
* Patient must be Eastern Cooperative Oncology Group (ECOG) performance status of = 2 and a life expectancy of more than 3 months.
* Patients must have adequate organ function.
* Patients must not have had prior surgery, chemotherapy, hormonal therapy, radiation therapy, or biological therapy for at least 4 weeks prior to starting study medication.
* Patients who were receiving mitomycin C, nitrosoureas, or carboplatin must be 6 weeks from the last administration of chemotherapy.
* Patients must not have an acute, critical illness,.
* All patients who are sexually active and able to conceive will be required to use contraception during treatment with lenalidomide

Design:

* A phase II trial in which patients are randomized to 2 dose levels of lenalidomide administered for 21 days every 28 days for 2 years.
* 76 patients (allowing for up to 3 inevaluable patients per dose level) will be enrolled over 4 to 5 years.
* The objective of the trial will be to determine in each of the two groups of patients (5 mg and 25 mg dose levels) whether, CC5013 is able to be associated with a response rate (partial response (PR) + complete response (CR)) that can rule out 10% (p0=0.10) in favor of an improved response rate of 30% (p1=0.30).

ELIGIBILITY:
-INCLUSION CRITERIA:

1. All patients with stage IV ocular melanoma, who have measurable disease will be considered.
2. Patients must have histopathological documentation of ocular melanoma confirmed in the Laboratory of Pathology/National Cancer Institute (NCI) of the Clinical Center at the National Institutes of Health. This can be from tissue obtained outside the National Institutes of Health (NIH).
3. Patient must be Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2.
4. Patients must have a life expectancy of more than 3 months.
5. Hematological eligibility parameters (prescreen):

   * Granulocyte count greater than 1,500/mm^3
   * Platelet count greater than 100,000/mm^3
   * If the creatinine is greater than 1.5 mg/dL, obtain a 24 hour urine collection. Creatinine clearance must be greater than 60 mL/min/1.73m^2.
   * Hepatic function: bilirubin (total) less than or equal to 2.0 mg/dl; Alanine aminotransferase (ALT) less than 10 x upper limit of normal; Aspartate aminotransferase (AST) less than 10 x upper limit of normal.
6. Patients must have recovered from any acute toxicity related to prior therapy or surgery, to a grade 1 or less unless specified above.
7. Patients must not have had prior surgery, chemotherapy, hormonal therapy, radiation therapy, or biological therapy, for at least 4 weeks prior to starting study medication. Patients who were receiving mitomycin C, nitrosoureas, or carboplatin must be 6 weeks from the last administration of chemotherapy.
8. Patients must not have an acute, critical illness, including a serious untreated infection.
9. Patients must be willing to return to the National Institutes of Health (NIH) for follow-up visits.
10. All patients who are sexually active and able to conceive will be required to use contraception during treatment with lenalidomide.

Only two criteria are allowed by the Food and Drug Administration (FDA) for the status of not of child bearing potential: hysterectomy or menopause for 24 consecutive months. Women of child bearing potential will be required to use two methods of birth control, one highly effective method and one additional method, at the same time during treatment and for one month after the completion of lenalidomide treatment. These methods must be used for at least four weeks before starting lenalidomide, during treatment, and for at least four weeks following the last dose of lenalidomide. Acceptable forms of birth control include:

Intrauterine device (IUD)

Latex condom

Hormonal (Birth control pills, injections, implants)

Diaphragm

Tubal Ligation

Cervical cap

Partner's vasectomy

Two barrier methods may be used if the physician agrees that the highly effective methods are medically contraindicated.

Women of childbearing potential must have a negative urine pregnancy test 24 hours prior to the start of lenalidomide.

Men who are sexually active must agree to use latex condoms.

Patients must be able to understand and sign informed consent form.

Patients must be greater than or equal to 18 years of age.

EXCLUSION CRITERIA:

1. Patients with evidence of active brain metastases will be excluded. Patients must have had a complete excision or radiotherapy and remain asymptomatic with stable disease as shown by magnetic resonance imaging (MRI) for at least six months.
2. Patients who are pregnant or lactating. No data is currently available about the excretion of lenalidomide in breast milk. Although no preclinical data suggest teratogenicity with this compound, because of the relationship to thalidomide, we will exclude patients who are pregnant or lactating.
3. Patients with a history of unstable or newly diagnosed angina pectoris, recent myocardial infarction (within 6 months of enrollment), New York class II-IV congestive heart failure, chronic obstructive lung disease requiring oxygen therapy or uncontrolled seizure activity are not eligible.
4. Patients who are known positive for human immunodeficiency virus (HIV) as it may increase their risk of infection since lenalidomide has effects on cells involved in the immune system.
5. Patients who have had prior therapy with lenalidomide.
6. Patients with known hypersensitivity reaction to lenalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caryn Steakley, Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gragoudas ES, Egan KM, Seddon JM, Glynn RJ, Walsh SM, Finn SM, Munzenrider JE, Spar MD. Survival of patients with metastases from uveal melanoma. Ophthalmology. 1991 Mar;98(3):383-9; discussion 390. doi: 10.1016/s0161-6420(91)32285-1. PMID 2023760
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/A_2005-C-0095.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 - 25 mg Lenalidomide (Revlimid) | Cohort 2 - 5 mg Lenalidomide (Revlimid)
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - 25 mg Lenalidomide (Revlimid) | Cohort 2 - 5 mg Lenalidomide (Revlimid) | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (7.6) | 58.86 (9.83) | 55.56 (9.71)
Gender [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 9 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Clinical Responses in Patients With Metastatic Ocular Melanoma
Description: Clinical response is assessed by the Response Evaluation Criteria for Adverse Events in Solid Tumors (RECIST). Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions. Progressive disease (PD) is at least a 20% increase in the sum of the LD of target lesions. Stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: 12 months
Population: Response data was combined for this outcome measure. Results are available for the combined cohorts only.
  Sixteen out of seventeen patients were eligible for response assessments.
Measure: Number; unit: Participants
Groups:
- Cohort 1 & 2 -25 mg & 5 mg Lenalidomide (Revlimid): oral dose (1 capsule) lenalidomide 25 mg per day 7 days a week for 3 weeks oral dose (1 capsule) lenalidomide 5 mg per day 7 days a week for 3 weeks
Arm/Group | Cohort 1 & 2 -25 mg & 5 mg Lenalidomide (Revlimid)
Number analyzed (Participants) | 16
Participants
  Complete Response | 0
  Partial Response | 0
  Progressive Disease | 9
  Stable Disease | 7

2. Primary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 24 months
Measure: Number; unit: Participants
Arm/Group | Cohort 1 - 25 mg Lenalidomide (Revlimid) | Cohort 2 - 5 mg Lenalidomide (Revlimid)
Number analyzed (Participants) | 8 | 9
Participants | 8 | 9

3. Secondary Outcome: Progression Free Survival
Description: Time interval from start of treatment to documented evidence of disease progression.
Time Frame: up to 2 years
Population: This outcome measure was not analyzed because the investigator left the institution.
Arm/Group | Cohort 1 & 2 -25 mg & 5 mg Lenalidomide (Revlimid)
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival
Description: Date of on-study to the date of death from any cause or last follow up.
Time Frame: up to 2 years
Population: This outcome measure was not analyzed because the investigator left the institution.
Arm/Group | Cohort 1 & 2 -25 mg & 5 mg Lenalidomide (Revlimid)
Number analyzed (Participants) | 0

5. Secondary Outcome: Determine Pharmacokinetics of Lenalidomide at Two Dose Levels: 5 mg and 25 mg
Description: Plasma samples will be obtained and plasma concentrations will be determined by a reversed-phase high-performance liquid chromatography (HPLC) assay using mass spectrometry (MS) detection.
Time Frame: Prior to treatment on cycle 1, day 1 and then on cycle 1, day 1 at 0.25, 0.5, 1, 2, 4, 6, 9 and 12 hours. Cycle 1, day 2 at 24 hours.
Population: This outcome measure was not analyzed because the investigator left the institution.
Arm/Group | Cohort 1 & 2 -25 mg & 5 mg Lenalidomide (Revlimid)
Number analyzed (Participants) | 0

6. Secondary Outcome: Determine Dose Level With Superior Efficacy and Acceptable Toxicity
Description: The most efficacious dose (with greater number of responses) with acceptable toxicity profile will be considered for use in subsequent trials. iI the number of responses is tied, then toxicity criteria (Common Terminology criteria (CTC) v3.0) will be used to select the preferred dose.
Time Frame: up to 2 years
Population: This outcome measure was not analyzed because the investigator left the institution.
Arm/Group | Cohort 1 & 2 -25 mg & 5 mg Lenalidomide (Revlimid)
Number analyzed (Participants) | 0

7. Secondary Outcome: Evaluate Effects of Lenalidomide on Pathways
Description: Tissue will be obtained to evaluate the effects of lenalidomide on pathways thought to be modulated by lenalidomide.
Time Frame: Baseline and at the end of treatment cycles 3 and 6. Every 21 day supply of lenalidomide with a 7 day rest (total of 28 days) will be considered a cycle of therapy.
Population: This outcome measure was not analyzed because the investigator left the institution.
Arm/Group | Cohort 1 & 2 -25 mg & 5 mg Lenalidomide (Revlimid)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Cohort 1 - 25 mg Lenalidomide (Revlimid) | Cohort 2 - 5 mg Lenalidomide (Revlimid)
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/9
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 25 mg Lenalidomide (Revlimid) (N=8) | Cohort 2 - 5 mg Lenalidomide (Revlimid) (N=9)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Death not associated with CTCAE term: Death Progression NOS (General disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 25 mg Lenalidomide (Revlimid) (N=8) | Cohort 2 - 5 mg Lenalidomide (Revlimid) (N=9)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 (2) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 2 (2) | 2 (3)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Alkaline phosphatase (Investigations) | 1 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (4) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 7 (14) | 3 (9)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2 (2) | 2 (5)
Flu-like symptoms (General disorders) | 1 (4) | 0 (0)
Hemoglobin (Investigations) | 3 (4) | 1 (1)
Infection with unknown ANC::Lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC::(Sinus) (Infections and infestations) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Musculoskeletal/Soft tissue - Other (Specify, tingling of hands and R foot) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (16) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 (3) | 1 (2)
Pain::Head/headache (Nervous system disorders) | 2 (2) | 1 (1)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain::Oral gums (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (3) | 2 (2)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vision-flashing lights/floaters (Eye disorders) | 1 (1) | 0 (0)
Bilirubin (hyperbilirubinemia) (Investigations) | 0 (0) | 1 (1)
Creatinine (Investigations) | 0 (0) | 1 (1)
hematoma (Vascular disorders) | 0 (0) | 1 (1)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 0 (0) | 1 (2)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (2) | 1 (2)
Leukocytes (total WBC) (Investigations) | 0 (0) | 1 (3)
Lymphopenia (Investigations) | 0 (0) | 1 (1)
Mood alteration::Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Pain: Back (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Pain: Extremity-limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No